CLINICAL TRIAL: NCT02528578
Title: Modulation of Painful Perception
Acronym: MODOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1208141; 2012-A01232-41 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2016-09

CONDITIONS: Healthy
Keywords: healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Device: thermal stimulation delivered by a thermode.; Other: functional MRI

INTERVENTIONS:
Device: thermal stimulation delivered by a thermode. — Empathetic context (neutral, empathetic, non-empathetic) when thermal stimulation
Other: functional MRI — MRI realised with thermal stimulations and empathetic context (neutral, empathetic, non-empathetic) when thermal stimulation

SUMMARY:
The objective of the study is to evaluate in healthy volunteers, the influence of empathy on pain perception.

It is widely accepted in the clinical management that the feeling of listening to the patients' pain would have a favorable influence on the pain, and conversely, the lack of listening would be aggravating.

In this study, the volunteer will receive painful thermal stimuli in empathetic context (l, empathetic or non-empathetic) Two situations will oppose, one where the examiner neglect or minimize the suffering of the voluntary and the other or the contrary, the subject will receive empathy.

The first part of the project is to verify that the pain is influenced by the empathetic context. The second part will be conducted functional MRI, which should isolate the brain regions affected by other people's empathy for pain.

ELIGIBILITY:
Inclusion Criteria:

* Right handed

Exclusion Criteria:

* Pregnant or lactating women,
* Against-indications to MRI
* Drug intake of less than 12 hours,
* Neurological history or deficits, psychiatric, auditory or visual.
* Decline to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Intensity of the perceived pain assessed by the volunteer by a analog scale (VAS) at each thermal stimulation. | Day 0

SECONDARY OUTCOMES:
blood-oxygen-level dependent (MRI) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (2):
- France (2):
  - Hospices Civils de LYON, Lyon
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No